CLINICAL TRIAL: NCT02962427
Title: Treatment of Post-dural Puncture Headache in Postpartum Parturients: Comparing Sphenopalatine Ganglion Block to Epidural Blood Patch.
Brief Title: Treatment of Post-dural Puncture Headache in Postpartum Patients: Sphenopalatine Ganglion Block to Epidural Blood Patch.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Decided to participate in a multicenter trial researching the same issue
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 16-1596
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Results first posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Sphenopalatine Ganglion Block; Blood Patch, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sphenopalatine Ganglion Block (Experimental): Sphenopalatine Ganglion Block: The patient is placed in the supine position. Four cc of 2% viscous lidocaine is placed to the level of the sphenopalatine ganglion with a 20 gauge angiocatheter along sterile swabs which were placed carefully into the patients nostrils bilaterally and lateral to the middle turbinate. It will be documented that the patient has no pain or paresthesia during or after the procedure. The swabs are withdrawn after 30 minutes.
  Interventions: Drug: Sphenopalatine ganglion Block
- Epidural blood patch (Active Comparator): Epidural Blood Patch: The patient is positioned in the sitting or lateral positon. Using aseptic technique, 20mL of autologous blood is drawn by a trained practitioner. The epidural placement is performed by a trained practitioner using aseptic technique and the vertebral space accessed is at or immediately below the original neuraxial placement. After entrance into the epidural space is confirmed with loss of resistance technique to either air or saline, 15-20 milliliters of sterile autologous venous blood is injected. After the procedure the patient rests supine for at least 1 hour. Patients are instructed to avoid heavy lifting, abdominal straining, or coughing for at least 48 hours.
  Interventions: Procedure: Epidural blood patch

INTERVENTIONS:
Drug: Sphenopalatine ganglion Block
  Other Names: SGB
  Arms: Sphenopalatine Ganglion Block
Procedure: Epidural blood patch
  Other Names: EBP
  Arms: Epidural blood patch

SUMMARY:
The purpose of this research study is to compare the effectiveness of a sphenopalatine ganglion block to an epidural blood patch for post-dural puncture headache relief in randomized postpartum parturients over a 48 hour period.

DETAILED DESCRIPTION:
The purpose of this research study is to compare the effectiveness of a sphenopalatine ganglion block to an epidural blood patch for post-dural puncture headache relief in randomized postpartum parturients over a 48 hour period. A known dural puncture is defined as free flow of cerebral spinal fluid (CSF) during neuraxial placement. An unknown dural puncture is defined as neuraxial placement where free flow of CSF is not appreciated, however the patient is diagnosed with a post-dural puncture headache as defined by the International Classification of Headache Disorders.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or age or greater
2. Postpartum obstetric parturient who was previously admitted to UCH.
3. Diagnosis of post-dural puncture headache based on the International Classification of Headache Disorders:

   1. Dural puncture has been performed
   2. Headache has developed within 5 days of the dural puncture
   3. Not better accounted for by another ICHD-3 diagnosis.
   4. Occurring immediately or within seconds of assuming an upright position and resolving quickly (within 1 minute) after lying horizontally.

Exclusion Criteria

1. Refusal to participate in the study
2. Placement of an EBP within the past 5 days
3. Allergy and/or intolerance to any the study materials
4. Contraindications to an EBP
5. Plan for therapeutic anticoagulation post-partum

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Wood, M.D., Principal Investigator — University of Colorado Anschutz Medical Campus - School of Medicine, Dept. of Anesthheisology
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Not sharing IPD with other researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- Sphenopalatine Ganglion Block: Sphenopalatine Ganglion Block: The patient is placed in the supine position. Four cc of 2% viscous lidocaine is placed to the level of the sphenopalatine ganglion with a 20 gauge angiocatheter along sterile swabs which were placed carefully into the patients nostrils bilaterally and lateral to the middle turbinate. It will be documented that the patient has no pain or paresthesia during or after the procedure. The swabs are withdrawn after 30 minutes.
  Sphenopalatine ganglion Block
- Epidural Blood Patch: Epidural Blood Patch: The patient is positioned in the sitting or lateral positon. Using aseptic technique, 20mL of autologous blood is drawn by a trained practitioner. The epidural placement is performed by a trained practitioner using aseptic technique and the vertebral space accessed is at or immediately below the original neuraxial placement. After entrance into the epidural space is confirmed with loss of resistance technique to either air or saline, 15-20 milliliters of sterile autologous venous blood is injected. After the procedure the patient rests supine for at least 1 hour. Patients are instructed to avoid heavy lifting, abdominal straining, or coughing for at least 48 hours.
  Epidural blood patch
Period: Overall Study
Arm/Group | Sphenopalatine Ganglion Block | Epidural Blood Patch
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sphenopalatine Ganglion Block | Epidural Blood Patch | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29 (4.36) | 30 (0) | 29.25 (3.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in The Numerical Rating Scale Pain Score
Description: The Numerical Rating Scale (NRS) is commonly used to evaluate pain level in patients. It is presented as a numerical scale of 11 options, numbered 0-10, where the patient's pain intensity is represented by a number between the extremes of 0 = no pain at all to 10 = worst pain imaginable in numerical fashion. Its simplicity, reliability, and validity have made the NRS a useful tool for describing pain severity or intensity. The Investigators will consider a difference of 20% as a clinically significant change in pain score.
Time Frame: Baseline and 48 hours
Population: Some subjects refused to give a 48 hour score.
Measure: Number; unit: score on a scale
Groups:
- Sphenopalatine Ganglion Block Baseline Score; Sphenopalatine Ganglion Block 48 Hours Score: Sphenopalatine Ganglion Block: The patient is placed in the supine position. Four cc of 2% viscous lidocaine is placed to the level of the sphenopalatine ganglion with a 20 gauge angiocatheter along sterile swabs which were placed carefully into the patients nostrils bilaterally and lateral to the middle turbinate. It will be documented that the patient has no pain or paresthesia during or after the procedure. The swabs are withdrawn after 30 minutes.
  Sphenopalatine ganglion Block
- Epidural Blood Patch Baseline Score; Epidural Blood Patch 48 Hours Score: Epidural Blood Patch: The patient is positioned in the sitting or lateral positon. Using aseptic technique, 20mL of autologous blood is drawn by a trained practitioner. The epidural placement is performed by a trained practitioner using aseptic technique and the vertebral space accessed is at or immediately below the original neuraxial placement. After entrance into the epidural space is confirmed with loss of resistance technique to either air or saline, 15-20 milliliters of sterile autologous venous blood is injected. After the procedure the patient rests supine for at least 1 hour. Patients are instructed to avoid heavy lifting, abdominal straining, or coughing for at least 48 hours.
  Epidural blood patch
Arm/Group | Sphenopalatine Ganglion Block Baseline Score | Sphenopalatine Ganglion Block 48 Hours Score | Epidural Blood Patch Baseline Score | Epidural Blood Patch 48 Hours Score
Number analyzed (Participants) | 3 | 2 | 1 | 1
score on a scale
  Subject 001: number analyzed (Participants) | 1 | 1 | 0 | 0
  Subject 001 | 8 | 0 |  |
  Subject 002: number analyzed (Participants) | 0 | 0 | 1 | 0
  Subject 002 |  |  | 8 |
  Subject 003: number analyzed (Participants) | 1 | 0 | 0 | 0
  Subject 003 | 4 |  |  |
  Subject 004: number analyzed (Participants) | 1 | 1 | 0 | 0
  Subject 004 | 10 | 5 |  |

ADVERSE EVENTS:
Time Frame: 48 hours
Description: Adverse events were collected during the 48 hour time period that participants were given either the sphenopalatine ganglion block or epidural blood patch
Arm/Group | Sphenopalatine Ganglion Block | Epidural Blood Patch
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT02962427/Prot_SAP_000.pdf